CLINICAL TRIAL: NCT06295055
Title: Evaluation of Clinical Outcomes of the Semi-rigid Shell Barrier System for Alveolar Bone Augmentation
Brief Title: Semi-rigid Shell Barrier System for Alveolar Bone Augmentation (SSBS for ABA)
Acronym: SSBS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Prisana Pripatnanont, Professor, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dentistry Prince of Songkla
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Guided Bone Regeneration; Bone Formation
Keywords: Guided bone regeneration; Bone augmentation; Semi-rigid shell; Semi-resorbable membrane

STUDY DESIGN:
Intervention Model Description: Before- after augmentation in patients with alveolar bone defects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- semi-rigid shell barrier system (Experimental): The semi-rigid shell barrier system is based on polycaprolactone (PCL) and biphasic calcium phosphate (BCP) in a 70:30 ratio.
  In vitro study, Tunthasen Pripatnanont et al. demonstrated that the semi-rigid shell barrier system exhibits suitable physical characteristics and mechanical properties, including appropriate morphology, hydrophilicity, adequate porosity, and a small pore size of less than 40 µm, facilitating angiogenesis and vascular penetration into the defect area. The semi-rigid shell demonstrates high resistance to compressive force, while the semi-resorbable covering membrane exhibits high elastic strength.
  In vivo studies have confirmed the effectiveness of the semi-rigid shell barrier system, showing bone and tissue integration after function, good stability, biocompatibility, and property as a barrier due to space-making and maintenance. The system also exhibits limited susceptibility to complications and ease of clinical handling during surgery.
  Interventions: Procedure: Ridge augmentation with semi-rigid shell barrier system

INTERVENTIONS:
Procedure: Ridge augmentation with semi-rigid shell barrier system — The semi-rigid shell, fixed to the outside cortex by tacks, acts as a bone wall. Bone particles are placed in the gap and covered with the semi-resorbable covering membrane, serving as a barrier membrane.

SUMMARY:
This study aims to compare the clinical outcome before and after augmentation in case series of 10 patients. The main question it aims to answer is Whether the semi-rigid shell system facilitates bone regeneration in moderate to severe alveolar bone defects after 4 months of bone augmentation. Participants with bone defects between 3 to 8 millimeters (moderate to severe bone defect) will be treated with xenograft covered with the semi-rigid shell barrier system as a stage approach technique for implant placement.

DETAILED DESCRIPTION:
Inclusion criteria are subjects requiring a bone defect between 3 to 8 millimeters (moderate to severe bone defect) covered 1-2 tooth span with adjacent tooth, planned for dental implant and fixed prosthesis, aged 20 and above but under the age of 65 with good physical health and good oral hygiene, able to comprehend and are willing to sign the consent form and can adhere to the protocol including scheduled clinic visits and assigned treatment and available for follow-up after implant placement.

Exclusion criteria are subjects in following reasons: (i) Heavy smokers (>10 cigarettes/day), (ii) receiving bisphosphonates, (iii) undergoing radiotherapy, (iv) uncontrolled medical conditions, (v) Alcoholism, (vi) Pregnancy Bone augmentation procedure Before surgery, patients will be premedication with 1000 mg of amoxicillin antibiotic and rinse chlorhexidine mouthwash 0.12% concentration for 1 minute. A single oral and maxillofacial surgeon will perform all surgical procedures. Local anesthesia with 4% Articaine hydrochloride with epinephrine 1: 100,000 (Septanest, Septodont, France) will be administered to each patient for inferior alveolar nerve block or local infiltration. A full thickness mucoperiosteal flap will be created, and the actual defect size will be measured with a periodontal probe following the flap procedure. Flap advancement with periosteal releasing flap, decorticate the bone with a round bur, then apply the semi-rigid shell and fix it with ti-tacks or screws. Following that, xenograft, a bone graft material will be placed, and ti-tacks will be used to fix the semi-resorbable covering membrane. Lastly, tension-free flap closure with double layer suturing technique which is a horizontal mattress and interrupts suture.

ELIGIBILITY:
Inclusion Criteria:

* subjects requiring a bone defect between 3 to 8 millimeters (moderate to severe bone defect) covered 1-2 tooth span with adjacent tooth
* Planned for dental implant and fixed prosthesis
* Aged 20 and above but under the age of 65 with good physical health and good oral hygiene
* Able to comprehend and are willing to sign the consent form and can adhere to the protocol including scheduled clinic visits and assigned treatment.
* Available for follow-up after implant placement.

Exclusion Criteria:

* (i) Heavy smokers (>10 cigarettes/day)
* (ii) receiving bisphosphonates
* (iii) undergoing radiotherapy
* (iv) uncontrolled medical conditions
* (v) Alcoholism
* (vi) Pregnancy.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Bone gain evaluation | 4 months
  CBCT images will be taken of the alveolar bone defect with an acrylic stent before the operation as a baseline, immediately post-operative, and 4 months after the operation. The most obvious point of the marker will be used to determine the vertical and horizontal bone gain.The distances from the reference points to the alveolar bone defect will be measured using analysis software.Any changes in the distances between the time points will be calculated in percentages.
Biocompatibility evaluation | 4 months
  The semi-resorbable covering membrane and the semi-rigid shell will be removed during the re-entry visit, and a trephine bone in size of 2x4 mm. will be analyzed using standard histology. The specimen will be fixed with 10% formalin, then the specimens will be embedded in paraffin, and longitudinal serial 5 μm-thick sections will be cut through their midline and stained with Hematoxylin and Eosin (H&E). The section slides will be scanned using a slide scanner (ScanScope, Aperio, USA) to create image files. The histological features of the specimens will be evaluated descriptively.

SECONDARY OUTCOMES:
Ridge volume change of alveolar ridge evaluation | 4 months
  The study will measure and analyze the volume change of the buccal alveolar ridge at baseline, 1 month, and 4 months after a bone augmentation procedure. The images will be obtained using an intraoral scanner and exported as stereolithography (STL) files. To minimize image distortion, matching and superimposition of 3D models of preoperative and postoperative bone defects will be conducted. The analysis of the data will be done using Geomagic Studio 1 software.The region of interest will be designated 10 mm. below the bone peak of adjacent teeth, and the volume of soft tissue in the targeted area will be calculated. The clinical ridge volume of bone defects will be measured in cubic mm. (mm.3) using a volumetric analysis tool.

CONTACTS AND LOCATIONS:
Overall Officials: Prisana Pripatnanont, Principal Investigator — Dentistry, Prince of Songkhla
Locations (1):
- Prince of Songkla, Songkhla, Hatyai, Thailand

IPD SHARING:
Plan to Share IPD: No